CLINICAL TRIAL: NCT05976724
Title: Investigation of the Effectiveness of Movement With Mobilization Technique for Distal Radial Fractures
Brief Title: Mobilization With Movement in Distal Radial Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, İSMAİL CEYLAN, Head of hand therapy clinic. PhD., Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12068451744
Record Dates: First submitted 2023-06-26; First posted 2023-08-04 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Pain; Acute Pain; Mobility Limitation
Keywords: Pain; Range of motion
MeSH Terms: conditions — Pain; Acute Pain; Mobility Limitation | interventions — Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Investigator and Outcomes Assessor are different people. The Outcome Assessor was blind to groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization with movement (Experimental): Mobilization with movement technique and traditional physiotherapy will be applied to the intervention group. Also patients will receive a traditional therapy program consisting of Conventional TENS and stretching and strengthening exercises.
  Interventions: Other: TENS, exercise; Other: Mulligan mobilisation
- Control group (Active Comparator): Patients will receive a traditional therapy program consisting of Conventional TENS and stretching and strengthening exercises.
  Interventions: Other: TENS, exercise

INTERVENTIONS:
Other: TENS, exercise — TENS: The patients were sat in a chair positioned next to a treatment table. The hand to be treated was placed on the treatment table with the forearm in the supine position. Electrodes were then placed on the transverse carpal ligament and palmar surface of the hand. Conventional TENS was applied, with the current transition time set to 50-100 µs, and performed at a frequency of 100 Hz for a period of 20 minutes at an amplitude that did not cause muscle contraction or any feeling of numbness or tingling.
  The supervised exercises were performed by the patients in a seated position. Strengthening exercises were performed with both hands by means of Digi-Flex hand exerciser (IMC Products Corp, Hicksville, New York), modeling mass and elastics. The patients were tasked with performing these exercises 10 times in each session and three times daily.
Other: Mulligan mobilisation — Each participant was tested with sustained manual glides in each of the possible directions during active wrist flexion and extension from the seated position. For the lateral glide, the therapist stabilises the lateral aspect of the distal radius using the first web-space. And glides the proximal row of carpal bones laterally (towards the thumb) using the first web-space of the other hand, following the joint line. For the medial glide, the therapist stabilises the medial aspect of the distal ulna using the first web-space. And glides the proximal row of carpal bones medially (away from the thumb) using the first web-space of the other hand, following the joint line.
  Arms: Mobilization with movement

SUMMARY:
Distal radius fractures (DRF) are the most common upper extremity disorders encountered in clinical practice. With an understanding of the mechanics of distal radius fractures, surgical intervention, and bone healing, the therapist can modify the therapy program according to the patient's individual needs. The therapeutic process is begun in the crucial stage of bone healing during fracture immobilization. By addressing edema reduction and early range of motion of the uninvolved joints, most problems can be avoided before cast or fixator removal. Rehabilitation following the immobilization period should focus on regaining wrist movements provided that earlier problems have been addressed properly. During the rehabilitative process, the therapist can incorporate scar management, modalities, joint mobilization, active and passive range of motion, splinting, and strengthening to maximize the patient's functional result.

Massage and mobilization techniques are used in the treatment of DRF due to their analgesic effects. The painless mobilization with movement technique (MWM, developed by Brian Mulligan) is a manual therapy method applies to correct the limitation of movement in the joint and to relieve pain and functional disorders. Many studies have shown that MWM technique provides faster and momentary painless joint movement compared to other physical therapy modalities. The patient group with DRF has a large place in the general population and long treatment processes cause both labour loss and economic loss. Therefore, this study aimed to examine the effectiveness of MWM technique in cases with distal radius fractures.

DETAILED DESCRIPTION:
In this study, 42 DRF patients with age range 18-65 who applied to Kırşehir Ahi Evran University Training and Research Hospital were examined. The individuals included in the study were divided into two groups according to the paired randomization method. These groups were control and intervention groups. Traditional physiotherapy methods were applied to the control group, traditional physiotherapy and MWM techniques were applied to the intervention group. Traditional physiotherapy methods were included; Transcutaneous Electrical Nerve Stimulation (TENS), stretching and strengthening exercises.

For the evaluation of patients; Visual Analogue Scale (VAS), wrist goniometric measurements, grip strength measurement, pinch strength measurement, edema measurement and Munich Wrist Questionnaire (MWQ) were used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with distal radius fracture

Exclusion Criteria:

* Patients with polytrauma,
* open fracture,
* ulnar head fracture (excluding ulnar styloid fracture),
* history of complex regional pain syndrome,
* limited cognitive capacity were excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 0-5 week
  Visual Analogue Scale (VAS). As a simple and commonly applied method, VAS is considered to be both valid and reliable in measuring patient pain intensity. The patients in the current study were each asked with indicating the intensity of their pain experienced within the past 24 hours by marking on a 10-cm line scale, where 0 = "No pain" and 10 = "Maximum pain

CONTACTS AND LOCATIONS:
Locations (1):
- İsmail Ceylan, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beselga C, Neto F, Alburquerque-Sendin F, Hall T, Oliveira-Campelo N. Immediate effects of hip mobilization with movement in patients with hip osteoarthritis: A randomised controlled trial. Man Ther. 2016 Apr;22:80-5. doi: 10.1016/j.math.2015.10.007. Epub 2015 Oct 31. PMID 26559319
- [Result] Cruz-Diaz D, Lomas Vega R, Osuna-Perez MC, Hita-Contreras F, Martinez-Amat A. Effects of joint mobilization on chronic ankle instability: a randomized controlled trial. Disabil Rehabil. 2015;37(7):601-10. doi: 10.3109/09638288.2014.935877. Epub 2014 Jul 3. PMID 24989067